CLINICAL TRIAL: NCT04597216
Title: Exploration of Feasability of Blood and Saliva Proteomic Analysis Through Harvesting by Silica Matrix
Brief Title: Exploration of Feasability of Blood and Saliva Proteomic Analysis Through Harvesting by Silica Matrix (NanoDx-CoV-19)
Acronym: NanoDxCoV19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC20.289
Record Dates: First submitted 2020-10-13; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: phase 1: patients with Covid-19 or with anotther respiratory infection phase 2 : patients with a supsected Covid-19
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unique arm (Other): there is only 1 arm in this study (all the participants will undergo the same diagnosis procedure)
  Interventions: Device: sample of blood and saliva

INTERVENTIONS:
Device: sample of blood and saliva — sample of 3ml of blood by veinous puncture, of 1 drop of blood by needlestick, and of saliva by spitting

SUMMARY:
Phase 1:

25 patients with a PCR-based diagnosis of Covid-19 will be be included to give 500 microliters of saliva and a 3 ml sample of blood for proteomic analysis; a drop of blood will also be put in a device connected to a silica matrix to perform spectrometric analyses. 25 patients with a non-Covid-19 respiratory infection will be included for the same samples. The proteomic analyses will be performed from classicaly draught blood, blood drop on silica, and saliva, to search for discriminating profiles between Covid-19 and non-Covid-19.

Phase 2:

150 patients with a suspected Covid-19 will be included at the same time than the Covid-19PCR is performed ; they will have a sample of saliva and of a drop of blood for proteomic analysis, whose results will be matched with PCR results.

DETAILED DESCRIPTION:
Phase 1: derivation analyses 25 patients with a PCR-based diagnosis of Covid-19 will be be included to give 500 microliters of saliva and a 3 ml sample of blood for proteomic analysis; a drop of blood will also be put in a device connected to a silica matrix to perform spectrometric analyses. 25 patients with a non-Covid-19 respiratory infection will be included for the same samples. The proteomic analyses will be performed from classicaly draught blood, blood drop on silica, and saliva, to search for discriminating profiles between Covid-19 and non-Covid-19.

Phase 2: confirmation analyses 150 patients with a suspected Covid-19 will be included at the same time than the Covid-19PCR is performed ; they will have a sample of saliva and of a drop of blood for proteomic analysis, whose results will be matched with PCR results.

ELIGIBILITY:
phase 1:

Inclusion Criteria for group 1:

* positive Covid-19 PCR
* clinical signs evocative of Covid-19

Exclusion Criteria for group 1:

* asymptomatic Covid-19 infection

Inclusion Criteria for group 1:

* negative Covid-19 PCR
* acute respiratory infection

Exclusion Criteria for group 1:

* none

Phase 2

Inclusion Criteria:

* suspicion of Covid-19
* sample for Covid-19 PCR planned or performed the same day
* admission ot emergency room exclusion criteria:
* past known Covid-19

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of proteomic profile | one day
  MALDI-TOF mass spectrometric analysis of blood and saliva proteins to obtain a specific proteomic profile (obtained or not)

SECONDARY OUTCOMES:
Interest of proteomic profile | one day
  Correlation between spectral analysis and severity of pathology at admission.
Stability of proteomic profile | two days
  Evaluation of mass spectrometric analysis reproductibility 48 hours after ambiant temperature conservation

CONTACTS AND LOCATIONS:
Locations (1):
- olivier EPAULARD, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided